CLINICAL TRIAL: NCT06513845
Title: Evaluating the Impact of Community-Based Mindfulness and Musical Programs on Psychiatric Measures, Drum Circle Synchrony Study 2c.a.
Brief Title: Drum Circle Synchrony Study 2c.a.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000028866_e; 2R25MH071584-11 (NIH)
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mental Health Issue; COVID-19
Keywords: Mindfulness; Meditation; Music
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Musicians group (Experimental): Musicians will listen to segments (~30 sec duration) of recordings taken from the music made during the previous drum circle and answer a survey asking how connected they felt while listening.Segments will be categorized as highly synchronized or not synchronized.
  Interventions: Behavioral: Communal drumming recordings
- Non-musicians group (Experimental): Non-musicians will listen to segments (~30 sec duration) of recordings taken from the music made during the previous drum circle and answer a survey asking how connected they felt while listening.Segments will be categorized as highly synchronized or not synchronized..
  Interventions: Behavioral: Communal drumming recordings

INTERVENTIONS:
Behavioral: Communal drumming recordings — Segments (~30 sec duration) of recordings taken from the music made during the previous drum circle. Segments will be categorized as highly synchronized

SUMMARY:
Mental health vulnerability due to stress is increased in People of African Descent (PADs) in America due to disproportionate effects of racism, poverty, education, and criminal justice sentencing. Various meditation and mindfulness approaches have provided evidence of measured reductions in multiple negative dimensions of stress. However, the majority of these studies do not have an adequate representation of PADs or other marginalized groups and are not designed to be culturally relevant or community based. Music has been shown to alleviate multiple symptoms of stress and has been shown to be a preferred and effective support for meditation and mindfulness. However, its role in stress management in PADs engaged in meditation or mindfulness is seldom studied. This study aims to evaluate the effects of a virtual, community-based music mindfulness program on stress management in PAD community members with anxiety and depression during COVID19.

2c.a. Drum Circle Synchrony Study: This study will investigate the role that synchrony plays in subjective feelings of connection.

DETAILED DESCRIPTION:
The investigators also propose a study to investigate the effects of communal drumming in reducing anxiety and increasing connectedness within drum circle community. Investigators hypothesize that these intervention will lead to reductions in scores on stress scales and will provide preliminary data for studies evaluating these types of community programs as an adjunct to the standard of care.

Musicians and non-musicians will listen to segments (~30 sec duration) of recordings taken from the music made during a previous arm of drum circle and answer a survey. Segments will be categorized as highly synchronized or not synchronized.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and older

Exclusion Criteria:

* ages 17 and younger

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Mean score connectedness rating | measured during listening session (30minutes)
  Mean connectedness rating survey assessed using a Likert scale total range of 1 (no connection) to 7 (maximum connection) for synchronous and asynchronous audio samples
Mean score subjective rating of synchrony | measured during listening session (30minutes)
  Subjective ratings of synchrony will be assessed using a Likert scale with total score range from 1-5, with higher scores indicating more synchrony, for synchronous and asynchronous audio samples.

CONTACTS AND LOCATIONS:
Overall Officials: AZA Allsop, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - BLOOM, New Haven, Connecticut
  - Musical Intervention Studios, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified, aggregate data will be shared through pre-prints, publications, and community town hall meetings.